CLINICAL TRIAL: NCT03197896
Title: A Neighborhood-Based Intervention to Reduce Prostate Cancer Disparities
Brief Title: Educational Intervention in Increasing Knowledge About Prostate Cancer in High-Risk Neighborhoods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15G.337
Record Dates: First submitted 2017-06-22; First posted 2017-06-23 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Prostate
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (prostate cancer information) (Experimental): The educator reviews general information about the prostate Cancer
  Interventions: Other: Educational Intervention
- Group II (general health information) (Active Comparator): The educator reviews topics about health promotion actions.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Review prostate cancer information

SUMMARY:
This clinical trial studies how well an educational intervention works in increasing knowledge about prostate cancer in high-risk neighborhoods. Learning about prostate cancer and the pros and cons of screening for prostate cancer may increase knowledge about prostate cancer while decreasing anxiety and concerns about prostate cancer screening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify neighborhoods with disproportionately high rates of advanced prostate cancer and describe patient- and neighborhood-level risk factors associated with the high-risk neighborhoods.

II. To develop, using a mixed methods approach, a targeted educational intervention about prostate cancer for men who live in high risk neighborhoods.

III. To test the impact of the targeted intervention on levels of knowledge, anxiety, and informed decision making about prostate cancer (PCa) screening.

IV. To observe the rates of PCa screening in the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Focus groups consisting of men who live, work, or worship in the 4 predetermined neighborhoods
* Currently reside in one of the four selected high risk neighborhoods

Exclusion Criteria:

• Men who do not reside in one of the four neighborhoods, who self-report that they have previously been diagnosed with prostate cancer, or who have had prostate cancer screening (prostatic specific antigen [PSA] or digital rectal examination [DRE]) within the past 12 months

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Themes identified by focus group transcripts | Up to 4 years
  Focus group transcripts will be analyzed by iterative rounds of coding by at least two members of the research team. Specific themes and trends will be identified within each transcript and discussed by the research team until final consensus is reached. Themes will be identified as topics that consistently occur across transcripts, as well as similarities and differences between transcripts.
Change in prostate cancer knowledge as measured by a 17-item scale | Baseline to up to 4 months
  Descriptive analyses will be used including t-test, frequency tables, nonparametric tests, correlations, regression models. Linear and generalized linear mixed models having random intercepts corresponding to neighborhood will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Charnita Zeigler-Johnson, MPH, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/